CLINICAL TRIAL: NCT06100315
Title: Nalbuphine as Adjuvant During Bilateral Suprazygomatic Maxillary Nerve Block for Pediatric Cleft Palate Repair: A Prospective, Randomized Comparative, Controlled Double-blind Study.
Brief Title: Nalbuphine as Adjuvant During Bilateral Suprazygomatic Maxillary Nerve Block for Pediatric Cleft Palate Repair
Status: Active, not recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reem Ayman Mahmoud, Principal Investigator, Assiut University
Other Study IDs: Nalbuphine in nerve block
Record Dates: First submitted 2023-10-14; First posted 2023-10-25 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Complication Following Peripheral Nerve Block
MeSH Terms: interventions — Nalbuphine; Bupivacaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bupivacaine: 30 patients will receive SMB using bupivacaine 0.125% of 0.2 ml/kg on each side (with maximum volume of 4 ml).
- Bupivacaine and Nalbuphine: 30 patients will receive SMB using bupivacaine 0.125 of 0.2 ml/kg + 0.1 mg/kg nalbuphine on each side (with maximum volume of 4 ml).
  Interventions: Drug: Nalbuphine

INTERVENTIONS:
Drug: Nalbuphine — bupivacaine 0.125% of 0.2 ml/kg and 0.1 mg/kg nalbuphine
  Other Names: Bupivacaine
  Groups: Bupivacaine and Nalbuphine

SUMMARY:
The aim of this study is to evaluate the efficacy of adding nalbuphine to bupivacaine via suprazygomatic nerve block for postoperative pain control and emergence agitation management in pediatrics aged from to 1 to 7 years who were maintained on sevoflurane inhalational anesthesia and scheduled for cleft lip and palate operation.

DETAILED DESCRIPTION:
Cleft lip and cleft palate are the most common craniofacial abnormalities in children. Cleft surgery results in a profound sympathetic stimulation leading to hypertension, tachycardia, and bleeding. Postoperative pain can be severe, and many of these patients are at increased risk of opioid-induced respiratory depression. Emergence agitation (EA) is another common problem in these children, with an incidence between 10% and 80% after sevoflurane anesthesia. Inadequate postoperative analgesia combined with vigorous crying may lead to surgical complications including wound dehiscence, bleeding, and respiratory compromise. The anesthetic management of cleft surgery should ideally bound the intraoperative autonomic response and provide adequate analgesia without respiratory depression or EA. A combination of inhalation-based anesthesia and high-dose opioids has been described to block the autonomic response during surgical dissection; however, this technique may be associated with postoperative sedation and respiratory depression. Surgical infiltration with a local anesthetic and a vasoconstrictor promotes hemostasis and reduces the autonomic response intraoperatively but does not provide extended postoperative pain relief. Sensory innervation of the lip and palate is provided by branches of the maxillary nerve. Suprazygomatic maxillary nerve blocks have been shown to be opioid-sparing after cleft lip and palate surgery. The addition of opioid analgesic might both prolong the analgesia after a regional nerve block and reduce the incidence of EA.

ELIGIBILITY:
Inclusion Criteria:

1. Age 1 to 7 years.
2. Both genders.
3. American society of anesthesiologists (ASA) physical state I-II.
4. Children undergoing palate surgeries.

Exclusion Criteria:

1. Guardians' refusal
2. History of developmental delay or mental retardation.
3. Children with any co-morbidities.
4. Skin infection at the site of injection.
5. Bleeding diathesis.
6. Known allergy to any drugs used in this study.

Ages: 12 Months to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Sample size calculation was carried out using G*Power 3 software. A calculated minimum sample of 54 pediatric patients will be needed and further randomly assigned into one of two equal groups (Group N - Nalbuphine group): 27 patients and Group B - Control arm): 27 patients, to detect an effect size of 0.5 in the mean value of postoperative pain control and emergence agitation management with an error probability of 0.05 and 80% power on a two-tailed test. But to avoid possible loss of samples (dropouts) during the study, the number of patients in each group will be increased to 30 to be a total of 60 patients.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
pain control | first day postoperative
  Postoperative pain will be assessed by FLACC which is (Face,Legs,Activity,Cry,Consolability) score in the first postoperative day.The scale is scored in the range of 0 - 10 with 0 representing no pain.10 representing severe pain. The scale has five criteria which are each assigned a score of 0, 1 or 2.

SECONDARY OUTCOMES:
Effect of nalbuphine with maxillary nerve block on postoperative emergence agitation according to WATCHA Scale "emergancy delirium scale" | first day postoperative
  The WATCHA scale is a four level arousal scale ranging from a "calm" patient (Score of 1) to "agitation with thrashing around" (Score of 4),"crying but can be consoled" is (Score of 2), "crying but cannot be consoled" is (Score of 3)
Asses the time for rescue analgesia | first day postoperative
  time to first dose of rescue analgesia, total amount of rescue analgesia in first 24 h postoperatively.
Asses the parents satisfaction | first day postoprrative
  Participants' satisfaction after the end of procedure the through 5-point Likert scale which is parent satisfaction score. (1 = very satisfied and willing to take the same medication and procedure in the future when indicated, 2 = satisfied, 3 = neither satisfied nor dissatisfied, 4 = dissatisfied, 5 = very dissatisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Ekram AA Osman, professor, Principal Investigator — Assiut University
Locations (1):
- Mohamed Fathy Mostafa, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Mostafa MF, Aal FAA, Ali IH, Ibrahim AK, Herdan R. Dexmedetomidine during suprazygomatic maxillary nerve block for pediatric cleft palate repair, randomized double-blind controlled study. Korean J Pain. 2020 Jan 1;33(1):81-89. doi: 10.3344/kjp.2020.33.1.81. PMID 31888322
- [Result] Mesnil M, Dadure C, Captier G, Raux O, Rochette A, Canaud N, Sauter M, Capdevila X. A new approach for peri-operative analgesia of cleft palate repair in infants: the bilateral suprazygomatic maxillary nerve block. Paediatr Anaesth. 2010 Apr;20(4):343-9. doi: 10.1111/j.1460-9592.2010.03262.x. Epub 2010 Feb 23. PMID 20199610